CLINICAL TRIAL: NCT02843321
Title: Combined Infusion of Cytotoxic T-Lymphocytes and Vaccination to Enhance Infection-Specific Immune Reconstitution Post-Allogeneic Stem Cell Transplantation
Brief Title: Combined Infusion of Cytotoxic T-Lymphocytes and Vaccination
Acronym: CYNTAX
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Responsible Party: Principal Investigator, David Gottlieb, Professor, University of Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cyntax
Record Dates: First submitted 2016-05-18; First posted 2016-07-25 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Complication of Transplant
Keywords: infection
MeSH Terms: conditions — Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T-cell infusion (Experimental): Infusion of donor-derived T cells. Non randomised, prevention study arm
  Interventions: Biological: T-cell infusion, influenza vaccination

INTERVENTIONS:
Biological: T-cell infusion, influenza vaccination — Donor derived infection-specific T-cells (with activity against CMV,adenovirus, EBV, VZV, Influenza, BKV and Aspergillus) and vaccination (with Fluvax)

SUMMARY:
To assess the safety and biological efficacy of prophylactically administered donor-derived multi-infection specific cytotoxic T lymphocytes (CTLs) (targeting cytomegalovirus (CMV), Adenovirus (Adv), Epstein Barr virus (EBV), Varicella-Zoster virus (VZV), Influenza (Flu), BK virus (BKV), and Aspergillus (Asp)) combined with early immunisation with Influenza and VZV vaccines for the prevention of viral and fungal infection following allogeneic blood or marrow stem cell transplantation.

DETAILED DESCRIPTION:
The study will analyse the safety and biological efficacy of administering the investigational products (donor-derived T cells stimulated with viral and fungal antigen expressing DC combined with Flu and VZV immunisation), for the prophylaxis of viral and fungal reactivation and/or infection following allogeneic blood or marrow transplantation. The cells will be given prophylactically a minimum of 28 days after transplantation followed by administration of the Flu and VZV vaccines 24 to 72 hours later. The AIMS are to study the safety of combining CTL infusions and vaccination as well as their effect on reconstitution of infection-specific immunity, viral and Aspergillus reactivation and infection rates after transplantation, viral load, and use of antiviral and antifungal pharmacotherapy for specific infections. The investigators will also evaluate the safety of infusions and vaccinations with respect to the development adverse events within the first 12 months post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing myeloablative or non-myeloablative allogeneic transplantation from an HLA (A, B and DR) identical or 1-3 antigen mismatched family or unrelated donor.
* Transplant performed for any type of non-malignant condition or haematological malignancy including but not limited to acute and chronic leukaemia, myelodysplasia, non Hodkgins and Hodgkin lymphoma or myeloma.
* Recipients of peripheral blood or bone marrow stem cells.
* Adequate hepatic and renal function (< 3 x upper limit of normal for AST (SGOT), ALT (SGPT), < 2 x upper limit of normal for total bilirubin, serum creatinine).
* Estimated life expectancy of at least 6 months.
* Patient (or legal representative) has given informed consent

Exclusion Criteria:

* Use of anti-lymphocyte globulin (ALG, ATG, Campath or other broad spectrum lymphocyte antibody) given in the 4 weeks immediately prior to infusion or planned within 4 weeks after infusion.
* Grade II or greater graft versus host disease within 1 week prior to infusion.
* Prednisone or methylprednisone at a dose of > 1 mg/kg (or equivalent in other steroid preparations) administered within 72 hours prior to cell infusion.
* Allergies to eggs or components of the Fluvax or Varivax vaccines.
* Privately insured in or outpatients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety of infection-specific T-cell infusion and vaccination | 1 week
  Presence of acute infusion related toxicities

SECONDARY OUTCOMES:
Change in infection specific immune reconstitution | 1 week, 2 weeks, 3 weeks, 4 weeks, 3 months, 6 months, 9 months, 12 months (post T-cell infusion)
Change in CMV, EBV and BKV load based on quantitive PCR | 1 week, 2 weeks, 3 weeks, 4 weeks, 3 months, 6 months, 9 months, 12 months (post T-cell infusion)
Use of specific anti-viral pharmacotherapy | 12 months (post T-cell infusion)
Use of systemic anti-fungal drugs including amphotericin and azoles | 12 months (post T-cell infusion)
Incidences of GVHD | 12 months (post T-cell infusion)
Number of in-hospital days following first discharge post transplant | 12 months (post T-cell infusion)

CONTACTS AND LOCATIONS:
Overall Officials: David Gottlieb, Professor, Principal Investigator — Westmead Hospital
Locations (1):
- Westmead Hospital Department of Haematology, Westmead, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No